CLINICAL TRIAL: NCT05604287
Title: A Placebo-controlled, Randomized, Double-blind, Single and Multiple Dose-escalation Study to Evaluate Safety, Tolerability, and Pharmacokinetics of ID119031166M With the Exploration of Pharmacodynamic Effects in Healthy Participants
Brief Title: Safety, Tolerability, and Pharmacokinetics of ID119031166M With the Exploration of Pharmacodynamic Effects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor have decided to cancel the trial
Sponsor: IlDong Pharmaceutical Co Ltd (Industry)
Collaborators: Parexel (Industry); YUNOVIA CO.,LTD. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ID119031166M-NASH-101
Record Dates: First submitted 2022-10-28; First posted 2022-11-03 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Healthy Participants
Keywords: First-in-human (FIH); Single ascending doses (SAD); Multiple ascending doses (MAD); Farnesoid X receptor (FXR) agonist; Noncirrhotic non-alcoholic steatohepatitis (NASH); Liver fibrosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- SAD: ID119031166M (Experimental)
  Interventions: Drug: ID119031166M
- MAD: ID119031166M (Experimental)
  Interventions: Drug: ID119031166M
- SAD: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- MAD: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ID119031166M — The participants will receive a single oral dose of ID119031166M or once daily oral doses of ID119031166M for 14 days.
  Arms: MAD: ID119031166M; SAD: ID119031166M
Drug: Placebo — The participant will receive a oral dose of Placebo.
  Arms: MAD: Placebo; SAD: Placebo

SUMMARY:
This study will evaluate safety, tolerability, and Pharmacokinetics (PK) of ID119031166M with the Exploration of Pharmacodynamic (PD) effects in Healthy Participants.

DETAILED DESCRIPTION:
This is a Phase 1, randomized, double-blind, placebo-controlled, sequential single/repeated-dose study. This study is a dose-escalation study with healthy participants in single ascending dose (SAD) including food-effect and multiple ascending dose (MAD) cohorts to determine the highest allowable dose (HAD).

ELIGIBILITY:
Inclusion Criteria:

* Must be Caucasian (White American of European or Latin American descent).
* Healthy participants of Japanese origin are allowed up to 50% in each MAD cohort.
* Body mass index (BMI) within the range of 18.5 to 30 kg/m^2 (inclusive) at the time of Screening.
* No congenital or chronic diseases that require treatment and without pathologic symptoms or signs on medical examinations.
* Participants with normal renal function.
* Women are eligible to participate if not pregnant, not breastfeeding. Male subjects should be willing to use 'highly effective' or 'applicable' contraceptive methods.

Exclusion Criteria:

* Currently have an acute disease with active symptoms.
* History of melanoma or other skin issues (including, but not limited to pre-cancerous areas, atopic dermatitis, psoriasis, rosacea, excessive moles etc.).
* History of clinically significant gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, psychiatric, musculoskeletal, or cardiovascular disease and/or arrhythmias.
* History of clinically significant hypersensitivity reaction to any drugs or additives.
* History of any gastrointestinal disease.
* History of substance use disorder including history of drug abuse disorder or history of alcohol use disorder, or tobacco use disorder or excessive caffeine intake.
* Evidence of moderate or excessive alcohol consumption.
* Tested positive in viral serology tests (hepatitis B virus [HBV], hepatitis C virus [HCV], and human immunodeficiency virus [HIV]).
* Known family history or known presence of long QT syndrome.
* A history of hypokalemia.
* Use of concomitant medicines that prolong QT/QTc (QT Interval Corrected for Heart Rate).
* History of active viral hepatitis (hepatitis A, B, C, and E), or autoimmune hepatitis.
* History of Multiple Endocrine Neoplasia type 2.
* Solid organ transplantation, except corneal transplants.
* History or presence of neutropenia which is defined as absolute neutrophil count (ANC) < 1.5 at Screening and admission.
* Participants with a microalbuminuria.
* Hemoglobin levels below 12.0 g/dL at Screening or Baseline.
* White Blood Cell levels below 3.5 × 109/L at Screening or Baseline.
* Platelet count < 150,000/µL, international normalized ratio (INR) > 1.5, albumin < 3.5 g/dL

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2024-04-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with Serious Adverse Events (SAEs) and Adverse Events (AEs) | From Screening (Day -28 to -3) until termination (approximately Day 8 for SAD and Day 22 for MAD)
  To evaluate the safety and tolerability of single and multiple ascending doses of ID119031166M in healthy participants.

SECONDARY OUTCOMES:
Maximum plasma concentration determined directly from the concentration- time profile (Cmax) | Day 1-4 for SAD and Day 1-17 for MAD
  To assess the PK of ID119031166M when given at single and multiple ascending doses in healthy participants.
  To explore food effect on PK of ID119031166M after a single-dose administration in healthy participants.
Time of maximum plasma concentration determined directly from the concentration-time profile (Tmax) | Day 1-4 for SAD and Day 1-17 for MAD
  To assess the PK of ID119031166M when given at single and multiple ascending doses in healthy participants.
  To explore food effect on PK of ID119031166M after a single-dose administration in healthy participants.
Area under curve from pre-dose (time 0) to the time of the last quantifiable concentration (tlast) (AUC0-last) | Day 1-4 for SAD and Day 1-17 for MAD
  To assess the PK of ID119031166M when given at single and multiple ascending doses in healthy participants.
Dose-normalized Cmax | Day 1-4 for SAD and Day 1-17 for MAD
  To assess the PK of ID119031166M when given at single and multiple ascending doses in healthy participants.
Dose-normalized AUC from pre-dose (time 0) extrapolated to 24 hours (AUC0-24) | Day 1-4 for SAD and Day 1-17 for MAD
  To assess the PK of ID119031166M when given at single and multiple ascending doses in healthy participants.
Dose-normalized AUC0-last | Day 1-4 for SAD and Day 1-17 for MAD
  To assess the PK of ID119031166M when given at single and multiple ascending doses in healthy participants.

CONTACTS AND LOCATIONS:
Locations (1):
- California Clinical trials medical group/PAREXEL, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: Undecided